CLINICAL TRIAL: NCT06503926
Title: Impact of COVID-19 Vaccination on Balance Function Among Adolescents: A Long-Term Perspective
Status: Completed | Type: Observational
Sponsor: Sinai University (Other)
Responsible Party: Principal Investigator, Alaa Noureldeen Kora, Lecturer, Sinai University
Other Study IDs: P.T.REC/012/005002
Record Dates: First submitted 2023-08-11; First posted 2024-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: SARS CoV 2 Vaccination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: SARS-COV-2 vaccination — Vaccination

SUMMARY:
Long term impact of COVID 19 vaccination on dizziness-related disability and balance in adolescence

ELIGIBILITY:
Inclusion Criteria:

* Adolescence age range 10-17
* received a dose or more of an approved COVID-19 vaccine at least one year before the study enrollment.

the ability to complete all assessment measures independently.

Exclusion Criteria:

1. vestibular or neurological disorders diagnosed before vaccination.
2. mixed COVID-19 vaccine types.
3. a history of traumatic brain injury.
4. current use of medications that affect balance.
5. documented COVID-19 infection within three months of assessment.
6. physical limitations that prevented them from completing balance testing.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: * Adolescence age range 10-17
  * Vaccinated by any available SARS -COV-2 Vaccinations
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-12-06 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Impact on Balance | Through study completion, an average of 1 day - 1 year after taking the vaccine
  The pediatric balance scale is used to assess balance (Lowest score =0 " worst"- Maximum score is 56 " Perfect Balance"
Functional Disability | Through study completion, an average of 1 day - 1 year after taking the vaccine
  The Dizziness Handicap Inventory is used to assess functional disability related to dizziness

SECONDARY OUTCOMES:
Emotional Disability | Through study completion, an average of 1 day - 1 year after taking the vaccine
  The Dizziness Handicap Inventory is used to assess emotional disability related to dizziness
Physical Disability | Through study completion, an average of 1 day - 1 year after taking the vaccine
  The Dizziness Handicap Inventory is used to assess physical disability related to dizziness

CONTACTS AND LOCATIONS:
Locations (1):
- Sinai University, Ismailia, Ismailia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No